CLINICAL TRIAL: NCT07025330
Title: A Phase IIa, Single-Site, Open-Label Study of Efgartigimod in Patients With IgG4-Related Disease
Brief Title: A Study of Efgartigimod in Patients With IgG4-Related Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Matthew C. Baker, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 79851
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: IgG4-related Disease
Keywords: efgartigimod; IgG4-RD; IgG4-related disease; FcRn; FcRn inhibitor
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- efgartigimod (Experimental): Participants will be treated with efgartigimod 1000 mg subcutaneously once weekly for up to 12 weeks
  Interventions: Drug: Efgartigimod

INTERVENTIONS:
Drug: Efgartigimod — efgartigimod 1000 mg subcutaneous injection given once weekly
  Other Names: efgartigimod alfa and hyaluronidase-qvfc

SUMMARY:
The goal of this clinical trial is to learn if efgartigimod can treat IgG4-related disease in adults. The main questions it aims to answer are:

In patients with IgG4-related disease, does treatment with efgartigimod reduce the volume of the:

* lacrimal gland(s) and/or
* salivary gland(s) and/or
* pancreas

Participants will:

* Receive efgartigimod once weekly for up to 12 weeks
* Visit the clinic every one to six weeks for checkups and tests
* Be asked to complete questionnaires to see how they feel on efgartigimod

ELIGIBILITY:
Key Inclusion Criteria:

* Have a clinical diagnosis of IgG4-related disease that requires treatment in the opinion of the investigator
* Meet the 2019 ACR/EULAR Classification Criteria for IgG4-Related Disease
* Have a serum IgG4 concentration greater than or equal to 2 times the upper limit of normal at Screening
* Have involvement of the lacrimal gland(s), salivary gland(s), and/or pancreas

  * If lacrimal and/or salivary glands are involved, it must be symptomatic, including but not limited to discomfort, pain, dryness, headache, or vision changes
  * If the pancreas is involved, it must be asymptomatic, diffuse enlargement without signs or symptoms of obstruction or evidence of major organ dysfunction in the opinion of the investigator
* Have a prior inadequate response to, or intolerance of, glucocorticoids, or who have experienced recurrent symptoms after previous treatment with glucocorticoids
* Are not receiving current treatment with immunosuppressive medications
* All women must test negative for pregnancy and agree to use a reliable method of birth control

Key Exclusion Criteria:

* Any exclusion criteria listed in the 2019 ACR/EULAR Classification Criteria for IgG4-Related Disease
* Prior treatment with an FcRn inhibitor
* Have conventional synthetic disease-modifying antirheumatic drug (csDMARD) or immunosuppressive use as follows:

  * Treatment with glucocorticoids within 28 days prior to Baseline or planned treatment during the study
  * Treatment with csDMARDs including but not limited to hydroxychloroquine, methotrexate, leflunomide, or sulfasalazine within 28 days prior to Baseline or planned treatment during the study
  * Treatment with cytotoxic or immunosuppressive drugs including but not limited to cyclophosphamide, mycophenolic acid, azathioprine, cyclosporine, sirolimus, or tacrolimus within 28 days prior to Baseline or planned treatment during the study
  * Treatment with a janus kinase (JAK) inhibitor including but not limited to tofacitinib, baricitinib, upadacitinib, or filgotinib within 28 days prior to Baseline or planned treatment during the study
  * Treatment with a Bruton's tyrosine kinase (BTK) inhibitor including but not limited to ibrutinib, zanubrutinib, acalabrutinib, pirtobrutinib, or rilzabrutinib within 28 days prior to Baseline or planned treatment during the study
* Have biologic disease-modifying antirheumatic drug (bDMARD) use as follows:

  * Treatment with etanercept, adalimumab, or anakinra within 28 days before Baseline or planned treatment during the study
  * Treatment with infliximab, certolizumab pegol, golimumab, abatacept, or tocilizumab within 56 days before Baseline or planned treatment during the study
  * Treatment with a B cell depleting agent including but not limited to rituximab, ocrelizumab, obinutuzumab, ofatumumab, inebilizumab, ianalumab, or obexelimab ≤ 6 months prior to Baseline
  * Patients who received B-cell targeted therapy > 6 and ≤ 12 months prior to Baseline must have a B-cell count that is within the laboratory reference range at Screening
  * Treatment with a BAFF antagonist including but not limited to belimumab or tabalumab within 6 months before Baseline or planned treatment during the study
  * Treatment with an IL-17 antagonist including but not limited to secukinumab, ixekizumab, or brodalumab within 6 months before Baseline or planned treatment during the study
  * Prior treatment with other bDMARDs may be allowed at the discretion of the investigator
* A history of, or current, inflammatory or autoimmune disease (that could affect the interpretation of safety or efficacy outcomes) other than IgG4-related disease
* Evidence of active tuberculosis, HIV, or hepatitis B or C infection
* History of cancer except for skin basal or squamous cell carcinoma, cervical dysplasia or carcinoma in situ that has been treated and is considered cured > 1 year prior to Baseline, prostate cancer considered cured for > 5 years with a normal prostate specific antigen, or colon cancer considered cured > 5 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in volume on FDG-PET/MRI of lacrimal gland(s) and/or | From Baseline to Week 12
Change in volume on FDG-PET/MRI of salivary gland(s) and/or | From Baseline to Week 12
  Salivary glands include parotid glands, submandibular glands, sublingual glands
Change in volume of pancreas on FDG-PET/MRI | From Baseline to Week 12

SECONDARY OUTCOMES:
Change in FDG avidity (SUVmax) of lacrimal glands on PET | Baseline to Week 12
Change in FDG avidity (SUVmean) of lacrimal glands on PET | Baseline to Week 12
Change in FDG avidity (total gland glycolysis) of lacrimal glands on PET | Baseline to Week 12
  Total gland glycolysis is SUVmean x gland volume
Change in FDG avidity (SUVmax) of salivary glands on PET | Baseline to Week 12
Change in FDG avidity (SUVmean) of salivary glands on PET | Baseline to Week 12
Change in FDG avidity (total gland glycolysis) of salivary glands on PET | Baseline to Week 12
  Total gland glycolysis is SUVmean x gland volume
Change in FDG avidity (SUVmax) of pancreas on PET | Baseline to Week 12
Change in FDG avidity (SUVmean) of pancreas on PET | Baseline to Week 12
Change in FDG avidity (total pancreatic glycolysis) of pancreas on PET | Baseline to Week 12
  Total pancreatic glycolysis is SUVmean x pancreatic volume
Change in exchange transfer (K^trans) of lacrimal glands on MRI | From Baseline to Week 12
Change in apparent diffusion coefficient (ADC) of lacrimal glands on MRI | From Baseline to Week 12
Change in microvascular volume fraction (f) of lacrimal glands on MRI | From Baseline to Week 12
Change in exchange transfer (K^trans) of salivary glands on MRI | From Baseline to Week 12
Change in apparent diffusion coefficient (ADC) of salivary glands on MRI | From Baseline to Week 12
Change in microvascular volume fraction (f) of salivary glands on MRI | From Baseline to Week 12
Change in apparent diffusion coefficient (ADC) of pancreas on MRI | From Baseline to Week 12
Change in T1 mapping of pancreas on MRI | From Baseline to Week 12
Change in T2 mapping of pancreas on MRI | From Baseline to Week 12
Change in extracellular volume (ECV) of pancreas on MRI | From Baseline to Week 12
Change in microvascular perfusion fraction of pancreas on MRI | From Baseline to Week 12
Change in serum IgG4 level | From Baseline to Week 12
Change in serum IgG level | From Baseline to Week 12
Change in serum IgE level | From Baseline to Week 12
Change in plasmablast count | From Baseline to Week 12
Change in absolute regulatory B cell count | From Baseline to Week 12
Change in IgG4-RD Responder Index | From Baseline to Week 12
Change in physician global assessment of disease | From Baseline to Week 12
  Symptoms rated on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state.
Change in patient global assessment of disease | From Baseline to Week 12
  Symptoms rated on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state.
Change in patient global assessment of ocular symptoms | From Baseline to Week 12
  Symptoms rated on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state.
Change in patient global assessment of salivary symptoms | From Baseline to Week 12
  Symptoms rated on a 100 mm VAS. Score range: 0 to 100, higher scores correspond to worse disease state.
Change in FACIT-F fatigue score | From Baseline to Week 12
  Total score range: 0-52, lower scores correspond with more fatigue.
Change in C3 laboratory assessment | From Baseline to Week 12
Change in C4 laboratory assessment | From Baseline to Week 12
Change in total IgG laboratory assessment | From Baseline to Week 12
Change in ESR laboratory assessment | From Baseline to Week 12
Change in CRP laboratory assessment | From Baseline to Week 12
Number of participants with safety endpoints of interest | From Screening to end of follow-up at Week 18
  Safety endpoints of interest include hypogammaglobulinemia, severe infection requiring hospitalization or IV antibiotics, and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C Baker, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No